CLINICAL TRIAL: NCT00676039
Title: Examination of the Pharmacokinetic Properties of Two Generic Antidepressants and Their Respective Brand Preparations in Healthy Male Volunteers
Brief Title: Comparison of the Pharmacokinetics of Two Generic Antidepressants and Their Respective Brand Preparations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Dr Pierre BLIER, University of Ottawa, Institute of Mental Health Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB-2007024
Record Dates: First submitted 2008-05-07; First posted 2008-05-12 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Healthy
Keywords: Therapeutic Equivalency; Human Experimentation; Bioequivalence; Brand name; Generic; Antidepressant; Healthy volunteers
MeSH Terms: interventions — Venlafaxine Hydrochloride; Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Crossover Effexor / NOVO-Venlafaxine
  Examination of the bioequivalence of Effexor (Wyeth Pharmaceuticals) and NOVO-Venlafaxine (NOVOPHARM).
  Both drugs will be given at the dose of 75 mg/day (one capsule per day) for 4 consecutive days. A washout period (corresponding to 10 half-life of the active metabolite desmethylvenlafaxine) will be respected after receiving each medication.
  Interventions: Drug: Venlafaxine; Drug: Effexor XR
- 2 (Active Comparator): Crossover Celexa/Gen-citalopram
  Examination of the bioequivalence of Celexa (Lundbeck, Brand Name) and Gen-Citalopram (Genpharm, Generic). Both drugs will be given at the dose of 40 mg/day (one tablet per day) for 8 consecutive days. A washout period (corresponding to 10 half-life of citalopram) will be respected after receiving each medication.
  Interventions: Drug: Gen-Citalopram; Drug: Celexa

INTERVENTIONS:
Drug: Venlafaxine — NOVO-Venlafaxine XR 75 mg (NOVOPHARM, Generic)
  Arms: 1
Drug: Gen-Citalopram — Gen-Citalopram 40 mg (Genpharm, Generic)
  Arms: 2
Drug: Effexor XR — Effexor XR 75 mg (Wyeth Pharmaceuticals, Brand Name)
  Arms: 1
Drug: Celexa — Celexa 40 mg (Lundbeck, Brand Name)
  Arms: 2

SUMMARY:
Generic medications should be the equivalent of brand medications with the exception of their price. Before a generic medication is introduced, its bioequivalence within a window of 80 to 125% of the original has to be demonstrated. There are reports that this criterion is not always followed in post-marketed periods. Such investigations were triggered by the observation that some patients previously stable on original medications relapsed when switched to a presumable equivalent generic. Several factors could account for this problem. Given reports of such problems occurring with the antidepressants citalopram and venlafaxine, some pharmacokinetic properties of specific brands of generics and the originals will be examined for these two medications. Twelve healthy male volunteers will participate in this crossover study. It is anticipated that there will be significant differences emerging between the two formulations given the clinical reports of patients deteriorating when switched from the original to the generic preparations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (absence of diseases: psychiatric, physical, neurological, metabolic,...)

Exclusion Criteria:

* Psychiatric disorder
* Hepatic disease
* Renal disease
* Gastrointestinal disease
* Hematological disease
* Smokers
* Physical and/or neurological disease
* Positive urine drug screen
* Abnormal blood pressure
* Abnormal urine/blood analysis (sodium, potassium, chloride, creatinine, urea, ALT, AST, total protein, glucose, and TSH)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Blood levels of drugs and their metabolite (when appropriate) will be evaluated for both the generic and the brand name medication. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Franck Chenu, Ph.D., Study Director — University of Ottawa
Locations (1):
- University of Ottawa, Institute of Mental Health Research, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Chenu F, Batten LA, Zernig G, Ladstaetter E, Hebert C, Blier P. Comparison of pharmacokinetic profiles of brand-name and generic formulations of citalopram and venlafaxine: a crossover study. J Clin Psychiatry. 2009 Jul;70(7):958-66. doi: 10.4088/jcp.09m05315. PMID 19653973